CLINICAL TRIAL: NCT01886092
Title: Verification of the Usefulness of the Repetitive Transcranial Magnetic Stimulation in the Treatment of Chronic Tinnitus
Brief Title: Repetitive Transcranial Magnetic Stimulation as a Treatment for Tinnitus
Acronym: rTMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-1212-081-451; SNUHT1 (Other: SNUHT1)
Record Dates: First submitted 2013-06-04; First posted 2013-06-25 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Tinnitus
Keywords: tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Active rTMS1 (Active Comparator): Combined low frequency frontal and temporal repetitive transcranial magnetic stimulation of left primary auditory cortex and left dorsolateral prefrontal cortex
  Interventions: Device: Active rTMS 1
- Active rTMS2 (Active Comparator): Temporal low frequency repetitive transcranial magnetic stimulation of left primary auditory cortex
  Interventions: Device: Active rTMS 2
- Active rTMS3 (Active Comparator): Frontal low frequency repetitive transcranial magnetic stimulation of left dorsolateral prefrontal cortex
  Interventions: Device: Active rTMS 3
- Sham Condition (Sham Comparator): Combined low frequency frontal and temporal repetitive transcranial magnetic stimulation of left primary auditory cortex and left dorsolateral prefrontal cortex
  Interventions: Device: sham condition

INTERVENTIONS:
Device: Active rTMS 1 — repetitive transcranial magnetic stimulation (Figured 8-Coil Cool-B65): 1000 stimuli of 1Hz rTMS over the left dorsolateral prefrontal cortex (110% motor threshold) followed by 2000 stimuli of 1 Hz rTMS over the left primary auditory cortex (110% motor threshold), each consisting of 4 days of rTMS treatment. (20 subjects).
  Arms: Active rTMS1
Device: Active rTMS 2 — repetitive transcranial magnetic stimulation (Figured 8-Coil MCF-B65): 3000 stimuli of 1 Hz rTMS over the left temporal cortex (110% motor threshold), each consisting of 4 days of rTMS treatment. (20 subjects)
  Arms: Active rTMS2
Device: Active rTMS 3 — repetitive transcranial magnetic stimulation (Figured 8-Coil MCF-B65): 3000 stimuli of 1 Hz rTMS over the left dorsolateral prefrontal cortex (110% motor threshold) each consisting of 4 days of rTMS treatment. (20 subjects)
  Arms: Active rTMS3
Device: sham condition — Sham rTMS, applied with the same combination of parameters as active rTMS, except for the number of stimulations per session. (20 subjects)
  Arms: Sham Condition

SUMMARY:
Efficacy of different protocols of transcranial magnetic stimulation for the treatment of tinnitus

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) of the dorsolateral prefrontal cortex has an add-on effect for primary auditory cortex rTMS in improving tinnitus-related distress. The investigators aimed to investigate whether rTMS of the dorsolateral prefrontal cortex and primary auditory cortex are capable of reducing tinnitus loudness.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic tinnitus
* Chronic subjective tinnitus for more than 6 months
* Subject is naive regarding rTMS
* Other concurrent treatments: A four-week washout from any other tinnitus treatment or management program is required prior to entering this study
* Stable enough to complete this study per the opinion of the Study Physician
* No restrictions, provided the dosages have been in place for at least 3 months
* A three month washout from any other tinnitus treatment or management program is required prior to entering this study.

Exclusion Criteria:

* Objective tinnitus or tinnitus with treatable cause
* Presence of intracranial or intraocular ferromagnetic materiel or particles
* Cardiac pacemaker or other electronic implants (including cochlear implant) Serious heart disease or other unstable major medical condition
* Personal history of central nervous system disorder, head injury, stroke or seizures
* Familial history of epilepsy
* Concomitant medication with antidepressants and antipsychotics
* Pregnant women
* Others known contraindications to rTMS or brain MRI

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-05; Primary Completion 2019-09 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Change of tinnitus severity as measured by the Tinnitus Handicap Inventory (THI) | Change from Baseline inTinnitus Handicap Inventory at 3 months

SECONDARY OUTCOMES:
Beck's Depression Inventory (BDI) | Baseline, before and after each intervention, 1, 2 and 3 months after the first intervention
State-Trait Anxiety Inventory (STAI) | Baseline, before and after each intervention, 1, 2 and 3 months after the first intervention
Pittsburgh Sleep Quality Index (PSQI) | Baseline, before and after each intervention, 1, 2 and 3 months after the first intervention
visual analogue scale (VAS) | Baseline, day 7, day 14, 1, 2 and 3 months after the first intervention

CONTACTS AND LOCATIONS:
Overall Officials: Myung-Whan Suh, MD, ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Noh TS, Kyong JS, Park MK, Lee JH, Oh SH, Suh MW. Dual-site rTMS is More Effective than Single-site rTMS in Tinnitus Patients: A Blinded Randomized Controlled Trial. Brain Topogr. 2020 Nov;33(6):767-775. doi: 10.1007/s10548-020-00797-y. Epub 2020 Sep 17. PMID 32944806
- [Derived] Noh TS, Kyong JS, Park MK, Lee JH, Oh SH, Chung CK, Kim JS, Suh MW. Treatment Outcome of Auditory and Frontal Dual-Site rTMS in Tinnitus Patients and Changes in Magnetoencephalographic Functional Connectivity after rTMS: Double-Blind Randomized Controlled Trial. Audiol Neurootol. 2019;24(6):293-298. doi: 10.1159/000503134. Epub 2019 Dec 12. PMID 31830753